CLINICAL TRIAL: NCT06322186
Title: Study to Actively Warm Trauma Patients-2 (STAYWARM-2): A Pilot Feasibility Trial of Chemical Versus Passive Warming Blankets in Massively Bleeding Patients
Brief Title: Study to Actively Warm Trauma Patients-2
Acronym: STAYWARM-2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STAYWARM-2 Trial
Record Dates: First submitted 2024-02-01; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2023-11

CONDITIONS: Trauma Injury; Hypothermia; Massive Hemorrhage
Keywords: Chemical heating blankets; Thermoregulation; Feasibility; Efficacy
MeSH Terms: conditions — Accidental Injuries; Hypothermia

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized 1:1 to receive either the experimental or control arm.
  Experimental arm: 2 Ready-Heat 4-panel blankets Control arm: standard of care (use of warmed blankets and forced air warmed blanket [FAWB])
Who Masked: Outcomes Assessor
Masking Description: Only the statistician will remain blinded during the final analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ready-Heat Blanket (Experimental): Two Ready-Heat 4-panel half blankets applied indirectly (as per manufacturer's directions) with two flannel blankets placed under them.
  Interventions: Other: Ready-Heat Chemical Heating Blankets
- Warmed blankets/FAWB (Active Comparator): Two warmed blankets (current standard of care) will be applied to the patient.
  Interventions: Other: Warmed blankets or FAWB

INTERVENTIONS:
Other: Ready-Heat Chemical Heating Blankets — Ready-Heat blankets are 4-panel half blankets that generate an oxygen-activated exothermic effect in 8-15 minutes (i.e., no electricity required), providing warmth over 8 hours at up to 40 degrees Celsius.
  Arms: Ready-Heat Blanket
Other: Warmed blankets or FAWB — The current standard of care for hypothermic patients is applying two warmed blankets or forced air warming blankets (FAWB).
  Arms: Warmed blankets/FAWB

SUMMARY:
Massively bleeding trauma patients have higher odds of mortality, increased hospital length of stay, and increased need for transfusion if they become hypothermic. Hypothermia is independently associated with mortality in traumatically injured patients due to its negative physiologic effects on hemostasis, cardiorespiratory and renal function.

Current warming strategies increase the logistical difficulty of transferring patients (which is frequent during the initial hours of trauma care) or must be changed at frequent intervals. Prehospital, military, and intraoperative studies have suggested chemical warming blankets as a pragmatic strategy to manage hypothermia. A recent pilot study (manuscript under review) at our institution demonstrated the feasibility of using the Ready-Heat® (TechTrade LLC, Orlando, FL, USA) chemical heating blanket in the initial phases of hospital care in bleeding trauma patients requiring a mass hemorrhage protocol (MHP). These self-warming blankets provide warmth over 8 hours at up to 40 degrees Celsius, carrying the advantage of portability with no continuous electric power requirement. Furthermore, the Ready-Heat blanket may be more effective than current strategies for rewarming patients at high risk of developing hypothermia. STAYWARM-2 will be the first randomized controlled trial performed in-hospital to evaluate a self-warming blanket to address hypothermia in massively bleeding trauma patients within the initial hours of hospital arrival.

This study will help to determine the efficacy and feasibility of using chemical heating blankets for hypothermia in the early hours of hospital care. This has potential to reduce the overall workload of direct care clinicians, freeing them for other patient care duties. Additionally, the intervention may achieve enhanced thermoregulation compared to current strategies, improving patient care and comfort, and avoiding the clinical complications related to hypothermia. Findings from this preliminary study may provide data for a future grant to launch a larger randomized controlled trial in the prehospital/in-hospital trauma setting to optimize the care of patients at risk of developing hypothermia.

DETAILED DESCRIPTION:
Patient screening, recruitment, and enrolment Recruitment will occur in the trauma bay during weekdays between 08:00-20:00hrs by Staff Trauma Team Leaders, with experience in QI initiatives and enrollment of severely bleeding trauma patients in clinical trials. Due to the high acuity of the patient condition, who usually needs multiple emergent interventions, consent will be obtained retrospectively (delayed consenting process). In addition, by seeking the patient's consent for enrollment during a tenuous point in their care, there is a potential of introducing bias, or concerns about coercion into accepting any care related to the initial resuscitation.

As soon as possible, following the randomization and inclusion, the patient (if able to comprehend) or substitute decision maker (SDM), will be approached about the study. They will have their specific warming intervention explained, and will have, at that point, the right to request that their data are withdrawn from the study.

Study personnel will contact the MRP for permission to approach the patient or ask that they introduce the study to the patient. With permission to enter the patient's circle of care, the research coordinator will then approach patients who were randomized and included in the study. The research coordinator will introduce the trial, confirm eligibility and conduct the informed consent discussion. This discussion will include the rationale for the study, the anticipated risks and benefits of participation, and their rights as a study participant (including withdrawal at any time). Capable participants will be offered an opportunity to ask questions and consult with their family and/or their physician before making a decision to continue in the study. If the patient is deemed incapable of providing informed consent for the study, study personnel will approach the SDM and go over the same process to obtain the consent. Patients or SDM will be given an Informed Consent Form to be signed, at this point.

One signed copy of the informed consent will be placed in the participant's medical record, another copy given to the participant and the original kept in the study file with the research coordinator. If the participant does not wish to participate, the reason for declining will be documented.

Patients will be randomized upon activation of the MHP according to a computer-generated allocation sequence using RedCap. If the patient is randomized to receive the intervention, the blood bank technologist will activate the two Ready-Heat® blankets by opening the seal on the packaging. The opened blankets will be attached outside of the first cooler of the MHP with red blood cells units sent to the trauma bay. The cooler will be transported by a porter, taken to the trauma bay and delivered to the trauma team. As this is an open-label trial, only the statistician will remain blinded during the final analysis. Enrollment will occur 08:00-20:00hrs on weekdays with the aim of assessing feasibility of using the blanket when study coordinators are not always available to reinforce temperature monitoring, proper blanket placement, and compliance with keeping the blanket on the patient over the intervention period.

Data will be collected by the research assistants and medical students as the patients are enrolled in the trial during weekdays 8 am to 8 pm. The Trauma Team Video Review Program, already implemented in the trauma bay, captures imaging and sound for all trauma resuscitations. The video review will permit granular data collection from admission to the trauma bay until the patient is transferred to the next phase of care. REDCap will be used to register the collected variables.

Research Ethics Board (REB) approval of the protocol and the informed consent form will be obtained. A recruitment log of eligible and ineligible patients as well as reasons for non-consent will be kept. We anticipate that this study will take 24 months to complete.

Storage and Stability As per manufacturer's Instructions for Use (IFU) document, the Ready-Heat® blanket may be stored in its air-tight protective packaging until ready for use. Upon removing the outer packing, the product will reach operating temperature within 15-20 minutes and will remain functional for up to 10 hours. After use, the blanket can be disposed of with regular waste as there are no harmful ingredients. The Blood Bank will maintain a stock of the Ready-Heat® blankets and stored at room temperature. The study product will be dispensed to those randomized to the intervention arm along with the first MHP pack of blood products.

Dispensing of Investigational Product The Ready-Heat® blanket will be provided to randomized patients by the Blood Bank along with the first MHP pack of blood products. An instruction sheet will be provided specifying how to apply the Ready-Heat blanket while avoiding direct skin contact. Instructions will be provided to keep the interventional products until the 8 hours post blanket application is completed.

Return and Destruction of Investigational Product Trauma Team members will be made aware of their responsibility to return any unused investigational products in the event the resuscitation is ended before applying the product (i.e.: patient death, termination of resuscitation). As per manufacturer's Instructions for Use (IFU) document, the Ready-Heat® blanket may be disposed of with regular waste as there are no harmful ingredients.

Study Visits and Assessments Study visits will be conducted by research assistants during weekdays to collect data

Study Visits

The following information will be collected during study visits either in person or remotely reviewing electronic health records and video recordings of patient resuscitations in the trauma bay. During weekdays, 8 am to 8 pm, the research assistant will be following the patient across the different phases/locations of care and will be collecting data at the same time. Video recordings will be performed as per Trauma Team Video Review policy for all patients. Video review will be used to assess time of blanket application in the Trauma Bay and reasons why the blanket was not applied or was removed. Research assistants will access all documented data and video recordings on the next weekday. Visits and specific data collection are detailed as follows:

Visit 1

On admission to the trauma bay: Demographics, injury characteristics and surgical management:

1. Date of injury
2. Time of injury
3. Sex
4. Age
5. Types of surgical procedures performed in the first 8 hours following hospital arrival
6. Date of arrival
7. Time of arrival
8. Time of randomization
9. Name of attending TTL and sub-TTL (if applicable)
10. Initial temperature recorded
11. Was the blanket placed on the patient? Yes/No
12. Time that the blanket was placed on the patient, if registered
13. Reason why blanket was not applied
14. Blanket applied directly to the patient's skin? Yes/No
15. Use of fluid warmers
16. Use of FAWB

Visit 2

Within the first eight hours of blanket application:

1. Location of the patient
2. Is the blanket kept on the patient? (Yes/No)
3. If not, what was the reason it was removed?
4. Temperature recorded, hourly (Yes/No)
5. If yes, the temperature recorded
6. Type of temperature measurement
7. Blanket applied directly to patient's skin? Yes/No
8. Use of FAWB
9. Use of fluid warmers

   At discretion of the clinician, within the first eight hours of blanket application:
10. Coagulation (platelet count, INR, fibrinogen)
11. Perfusion parameters (pH, base deficit, serum lactate)
12. Hemoglobin
13. Number of units of red blood cells, plasma, platelets, and fibrinogen concentrate administered within the first 8 hours

Visit 3

At 24 hours post blanket application:

1. Number of units of red blood cells, plasma, platelets, and fibrinogen concentrate administered within the first 24 hours
2. Type of injury (blunt/penetrating)
3. Injury Severity Score (ISS)
4. Frequency of safety events with skin

Compliance Monitoring and Assessment Throughout the study duration, compliance with application of the control or study intervention will be directly observed by research assistants on study visits, and retrospective review of video recordings in the trauma bay and the health records. The feasibility of adherence to temperature monitoring, and blood and serum monitoring as per clinician discretion will be evaluated. Any use of concurrent warming strategies (i.e.: fluid warmers, FAWB, etc.) will also be recorded.

Protocol Deviations Planned or unplanned deviations may occur on the part of the participant, the investigator, or study research team. In resolution to a deviation, corrective/preventative actions are to be developed and implemented in a timely manner to avoid subsequent deviations. Protocol deviations will be documented and reported as required and assessed where necessary during analysis. If a control or study intervention is noted to not be in use, or key data are missing from the health record, a reason for noncompliance will be documented. Based on findings from STAYWARM1, reasons for noncompliance are hypothesized to arise from patient condition, and lack of familiarity with the study protocol. Several educational initiatives will be developed prior to study commencement for trauma team members, to avoid protocol deviations during the study period.

ASSESSMENT OF SAFETY Definitions Adverse Event An Adverse Event (AE) is defined as any new event that may jeopardize the patient which the study investigator physician perceives may be directly related to the enrolment in the pilot study or to the assigned arm. Adverse events are not study related if they are related primarily to the underlying disease. All AEs are to be documented and assessed for relatedness. If related to the study intervention and occurring from baseline up to 24 hours (by the final visit), the AE will be recorded on the eCRF and coded as per the most recent edition of the Common Terminology Criteria for Adverse Events (CTCAE).

Expected adverse events with Ready-Heat® blankets Prolonged direct skin contact with the Ready-Heat blanket has been known to cause mild burns. The manufacturer specifies the need for careful supervision when used with "the elderly people with sensitive skin and those who can't feel heat or regulate heat"13. Given that some of the enrolled patients may be sedated due to clinical condition, the study products will be applied with the express direction to avoid direct skin contact. The recommendation will be made to use a standard blanket as an intermediary between the skin and the study product.

Unexpected Adverse Event An unexpected adverse event is defined as any adverse event that is not identified as expected or in nature, severity or frequency in the current Health Canada Product Monograph.

Serious Adverse Event (SAE)

A serious adverse event (SAE) in the study is defined as:

1. any event that is fatal or immediately life threatening, permanently disabling, severely incapacitating, or requires prolonged inpatient hospitalization, or
2. any event that may jeopardize the patient and requires medical or surgical intervention to prevent one of the outcomes listed above, AND
3. which the attending physician perceives may be directly related to enrolment in the study, or to the assigned arm.

   SAEs will be considered to be study-related if the event follows a reasonable temporal sequence from the study intervention and could readily have been produced by the intervention. Adverse events are not study related if they are related primarily to the underlying disease.

   Assessment of an Adverse Event Relationship (Causality/Relatedness) The causality assessment is the determination, according to the investigator's clinical judgment, of the existence of a reasonable possibility that the investigational product (IP) caused or contributed to an adverse event.

   If the investigator or delegated sub-investigator is unsure about whether or not the study product caused or is related to the event, then the event will be handled as "related" to the study product for reporting purposes of the trial. If the causality assessment is "unknown but not related" to the study product, this should be clearly documented in the source documents.

   Expectedness Events are classified as unforeseen or unexpected if the nature, severity, or frequency is not consistent with the risk information set out in Section 9.1.2 or the Product Monograph (PM) or label.

   Seriousness Events are classified as serious if associated with effects threatening the life or physiological functions of a participant. Refer to the definition for "Serious Adverse Events" in section 9.1.5.

   Severity The term "severe" is often used to describe the intensity (severity) of a specific event (e.g. mild, moderate, or severe myocardial infarction); the event itself, however, may be of relatively minor medical significance (such as severe headache). This is not the same as "serious," which is based on participant/event outcome or action criteria usually associated with events that pose a threat to a participant's life or functioning. The terms "serious" and "severe" are not synonymous. Seriousness (not severity) serves as a guide for defining regulatory reporting obligations.

   To assess the severity of an adverse event the investigators will use the following:

   ● the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE)

   Adverse Event Recording Investigations into potential adverse events should be done during each contact with a participant. Investigations may be done through specific questioning and, as appropriate, by examination. Information on all adverse events should be recorded promptly in the source document, and assessed by an investigator in a timely manner allowing sufficient time to meet required reporting timelines for SAEs and serious unexpected adverse drug reactions (SUADRs) if needed. Adverse event CRFs should be completed using source documents by a delegated research team member in a timely manner/within 15 days of site awareness. All clearly related signs, symptoms, and abnormal diagnostic procedures should be recorded in the source document, though should be grouped under one diagnosis. Each diagnosed adverse event should then be categorized in accordance with the revised NCI Common Terminology Criteria for Adverse Events (CTCAE).

   The following are not considered AEs and therefore do not require recording:
   * Pre-existing diseases or conditions identified and recorded at screening/baseline unless, at the discretion of the investigator, the disease or condition worsens in severity or frequency
   * At the discretion of the investigator, events considered likely manifestations of the underlying disease or that commonly occur in the study population independent of study drug exposure
   * Elective medical or surgical procedures.

   Procedures for Reporting a Serious Adverse Event and Unanticipated Events Investigator reporting: Notifying the REB Serious adverse events and unanticipated events should be recorded and reported to the REB in accordance with local reporting requirements and timelines.

   Investigator reporting: Notifying the Sponsor The investigator is responsible for reporting SAEs and SUADRs to the sponsor (Sunnybrook Research Institute) in accordance with applicable regulations and reporting requirements and timelines.

   Events that are assessed to be serious and unexpected and related or cannot be ruled out as related to the investigational product are considered SUADRs. Reporting for SUADRs should include a description of the event in sufficient detail to allow for a complete medical assessment of the case and independent determination of possible causality. The minimum information required includes at least one identifiable participant, one identifiable reporter, one serious reaction, and one suspect product.

   Additionally, for SAEs and SUADRS, a Suspect Adverse Reaction Report - CIOMS I Form (Appendix B) must be completed by the investigator and forwarded to the Sponsor within 24 hours of site awareness. Information on other possible causes of the event, such as concomitant medications and illnesses should also be provided as soon as is made available.

   Sponsor Reporting of SUADRs: Notifying Health Canada The regulatory sponsor is responsible for reporting SUADRs to regulatory authorities in accordance with local expedited reporting requirements and timelines. In addition, the Sponsor will complete the ADR Expedited Reporting Summary Form and submit this form in conjunction with the completed CIOMS Form to the appropriate Health Canada directorate.

   Sponsor Reporting of SUADRs: Notifying Sites The regulatory sponsor is responsible for distributing expedited reports of SUADRs to each investigator for submission to local Ethics Committees within 15 days of sponsor awareness.

   Reporting and Entry Timelines

   Study investigators will report SAEs to the sponsor within the following timelines:
   * All deaths and immediately life-threatening events, whether related or unrelated, will be recorded and reported to the sponsor within 24 hours of site awareness.
   * Serious adverse events other than death and immediately life-threatening events, regardless of relationship, will be reported to the sponsor within 72 hours of site awareness.

   Adverse event information will be entered into the CRF in a timely manner and no later than 15 days from the time the investigator becomes aware of the event.

   Serious adverse event information will be entered into the CRF in a timely manner/within 72 hours from the time the investigator becomes aware of the event.

   9.0 Early Termination and Reasons for Withdrawal

   While it is not anticipated to cause discomfort, patients may find that they are not able to continue with the study product due to the ongoing heat. Patients are permitted to withdraw consent at any time if they desire and will not undergo further trial investigations if they do so. Participants withdrawing from the study should be contacted by the study research team requesting a final visit and to follow up with any unresolved adverse events. Once withdrawn from the study, no further study procedures or evaluations should be performed, or additional study data collected. However, every effort should be made to obtain permission to document the reason for withdrawal and to collect participant outcomes, such as survival data up to the protocol-described end of participant follow up period, where possible. Any data collected prior to the withdrawal of consent may be retained and used by the sponsor. If the patient withdraws from the study, the research team will notify the patient's most responsible physician.

   Data Collection and Follow-up for Withdrawn Participants Patients will be asked to continue with follow-up of body temperature and laboratory tests. It is important to continue to follow these patients and capture outcomes that occur once they have discontinued study intervention to determine feasibility. Through telephone calls and emails, every effort will be made to obtain permission to document the reason participants withdrew consent and to continue collecting the body temperature and laboratory values previously mentioned. Patients who have had at least one of the blankets applied will be included in the per-protocol analysis.

   ETHICAL ISSUES Ethical conduct and ethical issues Approval for patient accrual must be obtained from research ethics board (REB) at SHSC before patient recruitment can begin. Any additional correspondence with REB must be maintained by the research coordinator/assistant.

   Informed Consent Due to the clinical condition of the patients during initial presentation, screening and enrollment will be at the discretion of the Trauma Team Leader on an urgent basis. When the patient is able to safely converse, study personnel will approach the Most Responsible Physician (MRP) for permission to approach the patient. With permission, the research coordinator will then approach enrolled patients, g to introduce the trial and conduct the informed consent discussion. By being invited into the patient's circle of care with the permission of the MRP, study personnel will Introduce the rationale for the study, the anticipated risks and benefits of participation, and their rights as a study participant (including withdrawal at any time). Capable participants will be offered an opportunity to ask questions and consult with their family and/or their physician before final decision. If the patient is deemed medically incapable, consent will be obtained from the substitute decision maker (SDM) . One signed copy of the informed consent will be placed in the participant's medical record, another copy given to the participant and the original kept in the study file with the research coordinator. If the participant does not wish to continue to participate, the reason for declining will be documented and the patient will be considered a screening failure (failure to provide informed consent).

   STUDY ADMINISTRATION This will be a single-site study, conducted at Sunnybrook Health Sciences Centre. The Research Coordinators, supervised by the Principal Investigator, will be responsible for trial coordination, site training, site start-up/activation, document management, supply management, database development, data management and statistical analysis. Study data and patient surveys will be entered and maintained on a secure password protected database developed using REDCap (www.projectredcap.org) and will be accessible via the Internet for data entry purposes.

   Arrangements for day-to-day management of the trial The research coordinator will be responsible for this aspect of the study, including system checks, maintenance, and data back-up. Patient data will be collected as enrollment occurs and entered into the electronic case report forms. Data queries will be generated monthly. A bi-weekly status report will include an update on the recruitment and status of all randomized patients. Monthly to bi-monthly audit and feedback meetings will be held. Protocol violations will be audited and recorded on designated Protocol Violation Forms. Clinical research coordinators will work with investigators on start-up activities (REB applications; study contract; organizing study materials; local in-services). Thereafter, research coordinators will screen, consent, and enroll patients, complete case report forms, and respond to data queries.

   Quality Assurance Study data will be maintained on a secure password protected database accessible from the world-wide-web. Quality control will be ensured by oversight by the research coordinator at Sunnybrook Research Institute, who will review the electronic data for all participants on a regular basis for completeness and consistency.

   Quality and completeness of data entry will be reviewed as soon as possible after data entry, within five business days of data entry for the first five participants randomized, and within 15 days of data entry thereafter. Data queries generated by identification of incomplete or inconsistent data will be raised and should be resolved by the study coordinator or PI in a timely manner. Corrections or changes in the data management system are tracked with the retention of the original data and the corrected data with the date of data entry and submitting personnel

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 16 years
* Requires massive hemorrhage protocol activation in the trauma bay
* Admitted to the trauma bay between 08:00-20:00 on a weekday

Exclusion Criteria:

* Transferred from another healthcare facility
* Death in the trauma bay prior to randomization
* Arrival to trauma bay with ongoing CPR
* Patients with penetrating head injury with Glasgow Coma Scale of 3 and loss of brain matter through the wound

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
An increase of 1⁰C at eight hours from the time of blanket placement | 0-8 hours from trauma bay arrival/blanket application
  To evaluate the effectiveness of the Ready-Heat® blanket to increase temperature by at least 1⁰C at eight hours from the time of blanket placement in the trauma bay in severely injured trauma patients who required massive hemorrhage protocol activation.
  Temperature will be measured upon arrival to the trauma bay and at 8 hours from arrival to trauma bay/time of blanket application.
Adherence to the 2 blankets application in the trauma bay in at least 80% of patients. | 0-90minutes (from trauma bay arrival until the patient leaves the trauma bay to the next phase of care - generally 30 to 90 minutes from arrival).
  Adherence to the application of the 2 Ready-Heat® blankets in patients enrolled in the intervention arm throughout the trauma bay resuscitation.
  Research personnel will record whether the 2 blankets were applied remained on the patient in the trauma bay.
Adherence to body temperature measurements (in degrees Celsius) 80% of each of the phases of initial care up to 8 hours following admission. | 0-8 hours from trauma bay arrival/blanket application
  Feasibility of body temperature measurement throughout the different phases of care (i.e.: TB, ED, CT scanner suite, OR, IR suite, ICU) within the first eight hours of blanket application. The temperature will be mesured on arrival to the trauma bay, prior to leaving the trauma bay, prior to leaving the CT scanner suite, prior to leaving the ED to the OR or IR, prior to leaving the IR suite, in the OR as per anesthesia standards, on arrival to the ICU, and at 8 hours time point (time point when the blanket will be removed) or the time point when the patient's temperature reaches 37.0 degrees Celsius.
  Research personnel will request/record temperature measurements at the time of trauma bay arrival and at any subsequent phases of care up to eight hours from blanket application.
Adherence to maintain the blankets applied on the patient in 80% of each of the phases of initial care up to 8 hours following admission. | 0-8 hours from trauma bay arrival/blanket application
  Feasibility of maintaining at least one blanket applied throughout the different phases of care (i.e.: TB, ED, CT scanner suite, OR, IR suite, ICU).
  Research personnel will monitor and record whether the 2 blankets remained on the patient throughout the phases of care.

SECONDARY OUTCOMES:
Concurrent warming strategies | 0-8 hours from trauma bay arrival/blanket application
  Concurrent warming strategies used (i.e.: fluid warmers, FAWB, etc.) within the first eight hours of admission/blanket application in conjunction with or replacement of Ready-Heat® chemical heating blanket.
Blood product usage | Within 24 hours post-blanket application/admission.
  Number of units of blood products (plasma, red blood cells, platelets, fibrinogen concentrate) transfused within 24 hours of trauma bay arrival
Coagulation parameter 1: platelet count | 0-24 hours from trauma bay arrival/blanket application
  platelet count (x10^9) will be recorded on arrival to the trauma bay and at the next time points as per clinician discretion, up to 24 hours following admission.
Coagulation parameter 2: INR | 0-24 hours from trauma bay arrival/blanket application
  International Normalized Ratio (INR) will be recorded on arrival to the trauma bay and at the next time points as per clinician discretion, up to 24 hours following admission.
Coagulation parameter 3: fibrinogen | 0-24 hours from trauma bay arrival/blanket application
  Fibrinogen (g/L) will be recorded on arrival to the trauma bay and at the next time points as per clinician discretion, up to 24 hours following admission.
Perfusion parameter 1: pH | 0-24 hours from trauma bay arrival/blanket application
  pH will be recorded on arrival to the trauma bay and at the next time points as per clinician discretion, up to 24 hours following admission.
Perfusion parameter 2: base deficit | 0-24 hours from trauma bay arrival/blanket application
  Base deficit (mmol/L) will be recorded on arrival to the trauma bay and at the next time points as per clinician discretion, up to 24 hours following admission.
Perfusion parameter 3: serum lactate | 0-24 hours from trauma bay arrival/blanket application
  Serum lactate (mmol/L) will be recorded on arrival to the trauma bay and at the next time points as per clinician discretion, up to 24 hours following admission.
Hemoglobin level | 0-24 hours from trauma bay arrival/blanket application
  Hemoglobin level measured on arrival, and at the next time points collected as per clinician discretion, up to 24 hours following admission.
Blanket placed directly on skin | 0-8 hours from trauma bay arrival/blanket application
  Number of times the Ready-Heat chemical heating blanket(s) are placed on the skin directly (without regular blankets underneath). Safety measure 1.
Skin redness and/or burns | 0 - 24 hours post-blanket application
  Number of times skin redness and/or burns occurs due to blanket application. Safety measure 2.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Da Luz, MD, Principal Investigator — Sunnybrook Health Sciences Centre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reynolds BR, Forsythe RM, Harbrecht BG, Cuschieri J, Minei JP, Maier RV, Moore EE, Billiar EE, Peitzman AB, Sperry JL; Inflammation and Host Response to Injury Investigators. Hypothermia in massive transfusion: have we been paying enough attention to it? J Trauma Acute Care Surg. 2012 Aug;73(2):486-91. PMID 23019675
- [Background] Dirkmann D, Hanke AA, Gorlinger K, Peters J. Hypothermia and acidosis synergistically impair coagulation in human whole blood. Anesth Analg. 2008 Jun;106(6):1627-32. doi: 10.1213/ane.0b013e31817340ad. PMID 18499589
- [Background] Lester ELW, Fox EE, Holcomb JB, Brasel KJ, Bulger EM, Cohen MJ, Cotton BA, Fabian TC, Kerby JD, O'Keefe T, Rizoli SB, Scalea TM, Schreiber MA, Inaba K; PROPPR study group. The impact of hypothermia on outcomes in massively transfused patients. J Trauma Acute Care Surg. 2019 Mar;86(3):458-463. doi: 10.1097/TA.0000000000002144. PMID 30444856
- [Background] Perlman R, Callum J, Laflamme C, Tien H, Nascimento B, Beckett A, Alam A. A recommended early goal-directed management guideline for the prevention of hypothermia-related transfusion, morbidity, and mortality in severely injured trauma patients. Crit Care. 2016 Apr 20;20(1):107. doi: 10.1186/s13054-016-1271-z. PMID 27095272
- [Background] Rajagopalan S, Mascha E, Na J, Sessler DI. The effects of mild perioperative hypothermia on blood loss and transfusion requirement. Anesthesiology. 2008 Jan;108(1):71-7. doi: 10.1097/01.anes.0000296719.73450.52. PMID 18156884
- [Background] Frank SM, Fleisher LA, Breslow MJ, Higgins MS, Olson KF, Kelly S, Beattie C. Perioperative maintenance of normothermia reduces the incidence of morbid cardiac events. A randomized clinical trial. JAMA. 1997 Apr 9;277(14):1127-34. PMID 9087467
- [Background] Slotman GJ, Jed EH, Burchard KW. Adverse effects of hypothermia in postoperative patients. Am J Surg. 1985 Apr;149(4):495-501. doi: 10.1016/s0002-9610(85)80046-5. PMID 3985289
- [Background] Phillips D, Bowman J, Zafren K. Successful Field Rewarming of a Patient with Apparent Moderate Hypothermia Using a Hypothermia Wrap and a Chemical Heat Blanket. Wilderness Environ Med. 2019 Jun;30(2):199-202. doi: 10.1016/j.wem.2019.01.001. Epub 2019 Feb 26. PMID 30824366
- [Background] Bennett BL, Holcomb JB. Battlefield Trauma-Induced Hypothermia: Transitioning the Preferred Method of Casualty Rewarming. Wilderness Environ Med. 2017 Jun;28(2S):S82-S89. doi: 10.1016/j.wem.2017.03.010. Epub 2017 May 5. PMID 28483389
- [Background] Oden TN, Doruker NC, Korkmaz FD. Compliance of Health Professionals for Prevention of Inadvertent Perioperative Hypothermia in Adult Patients: A Review. AANA J. 2022 Aug;90(4):281-287. PMID 35943754
- [Background] Munday J, Delaforce A, Forbes G, Keogh S. Barriers and enablers to the implementation of perioperative hypothermia prevention practices from the perspectives of the multidisciplinary team: a qualitative study using the Theoretical Domains Framework. J Multidiscip Healthc. 2019 May 29;12:395-417. doi: 10.2147/JMDH.S209687. eCollection 2019. PMID 31239694
- [Background] Torossian A, Van Gerven E, Geertsen K, Horn B, Van de Velde M, Raeder J. Active perioperative patient warming using a self-warming blanket (BARRIER EasyWarm) is superior to passive thermal insulation: a multinational, multicenter, randomized trial. J Clin Anesth. 2016 Nov;34:547-54. doi: 10.1016/j.jclinane.2016.06.030. Epub 2016 Jul 17. PMID 27687449
- [Background] Khayyat H, Callum JL, Hill-Strathy M, Strauss R, Notario L, Nathens A, da Luz L. Compliance with the massive hemorrhage protocol in trauma: a retrospective quality review. Can J Anaesth. 2021 Jan;68(1):156-158. doi: 10.1007/s12630-020-01806-1. Epub 2020 Sep 16. No abstract available. PMID 32936441
- [Background] Callum JL, Yeh CH, Petrosoniak A, McVey MJ, Cope S, Thompson T, Chin V, Karkouti K, Nathens AB, Murto K, Beno S, Pendergrast J, McDonald A, MacDonald R, Adhikari NKJ, Alam A, Arnold D, Barratt L, Beckett A, Brenneman S, Chaudhry HR, Collins A, Harvey M, Lampron J, Margarido C, McFarlan A, Nascimento B, Owens W, Pai M, Rizoli S, Ruijs T, Skeate R, Skelton T, Sholzberg M, Syer K, Viveiros JL, Theriault J, Tinmouth A, Van Heest R, White S, Zeller M, Pavenski K. A regional massive hemorrhage protocol developed through a modified Delphi technique. CMAJ Open. 2019 Sep 3;7(3):E546-E561. doi: 10.9778/cmajo.20190042. Print 2019 Jul-Sep. PMID 31484650
- See also: Ready-Heat Blanket Product Website — https://www.ready-heat.com

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT06322186/Prot_SAP_000.pdf